CLINICAL TRIAL: NCT00738608
Title: Etoricoxib as a Pre-emptive Analgesic in Therapeutic Arthroscopy
Status: Completed | Type: Observational
Sponsor: Marienkrankenhaus Soest (Other)
Responsible Party: Dr. Lierz, Marienkrankenhaus Soest
Other Study IDs: 2006-000451-17
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Pain
Keywords: morphine; consumption; postoperative; pain; Pain during 24h postoperative; Morphine consumption in 24h postoperative
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 33 pat. with verum
- 2: 33 Pat. with placebo

SUMMARY:
The aim of this study is to demonstrate that compared to placebo the preoperative administration of a single dose of 120 mg etoricoxib can provide adequate pain relief in the postoperative phase while reducing the need for systemic opioids. The primary endpoint is the decrease of systemic opioid use.

DETAILED DESCRIPTION:
Depending on the pain intensity, various analgesics are used in the prevention of surgical wound pain. For severe pain, opioids like piritramide and morphine are used. These can be given at fixed intervals, continuously, as required or by patient-controlled analgesia (PCA). The method used depends on the equipment and supervision available and on the patient's cooperation. However, with all the methods of administration mentioned there is a risk of respiratory depression because strong opioids are used. Weak opioids like tramadol can be given as alternatives to piritramide and morphine, a combination of tramadol and metamizol having proven effective. Often an antiemetic is given as well, as many patients who receive the combination experience nausea and vomiting. For mild pain metamizol or a nonsteroidal anti-inflammatory drug (NSAID) is often sufficient on its own.

As some controversy is attached to the use of metamizol because of the risk of agranulocytosis (metamizol was withdrawn from the Scandinavian market in 1999), some hospitals do not use the drug. The use of NSAIDs is likewise problematic. They can cause, for example, gastric ulcers in predisposed patients. In the setting of the stress accompanying surgery, however, even previously unremarkable patients can quickly develop stress ulcers. Another problem with NSAIDs is that they affect blood clotting to various extents by inhibiting platelet aggregation. This aspect is particularly crucial in the early treatment of postoperative pain when intact blood clotting is essential. An ideal analgesic for postoperative pain would not induce respiratory depression nor affect blood clotting nor cause gastric ulcers. Because inhibiting the enzyme cyclooxygenase-1 (COX-1) increases the effects on the gastric mucosa and on platelet aggregation, an analgesic should selectively inhibit only the enzyme cyclooxygenase-2 (COX-2), which mediates inflammatory processes. This is the rationale behind using COX-2 inhibitors in the treatment of acute pain. With selective COX-2-inhibiting analgesics it is possible to inhibit inflammatory processes without favoring the occurrence of clotting disturbances or gastric mucosal lesions. Such an analgesic is available in the form of etoricoxib, which exhibits greater COX-2 selectivity than other coxibs so far approved. Etoricoxib has mainly been used for the treatment of pain associated with osteoarthritis and rheumatoid arthritis pain and for chronic pain (lower back pain). However, coxibs have also been used with impressive results in the treatment of acute peri- and postoperative pain. Thus, a 50 mg preoperative dose of rofecoxib not only significantly decreased the postoperative need for analgesics but also reduced postoperative pain.

Etoricoxib exhibits similar properties to rofecoxib. It is already approved for the treatment of acute pain in Australia, Latin America (except Argentina), Mexico, Hong Kong, Singapore, Malaysia, the Philippines, Thailand, and Indonesia. The preoperative use of Etoricoxib could provide reliable analgesia in the postoperative phase with a potency comparable to that of NSAIDs and other coxibs but without affecting blood clotting processes or favoring the occurrence of gastric ulcers

ELIGIBILITY:
Inclusion Criteria:

* Knee arthroscopy

Exclusion Criteria:

* Opiate addiction
* Pregnancy or breast-feeding
* Known hypersensitivity to the active substance or to any of the excipients of the film tablet
* Active peptic ulcer or active gastrointestinal bleeding, inflammatory bowel disease, severe hepatic dysfunction (serum albumin <25 g/l or Child-Pugh score ≥10).
* Further exclusion criteria are congestive heart failure (NYHA II-IV), hypertension with not adequately controlled blood pressure, established ischemic heart disease, peripheral arterial disease, and/or cerebrovascular disease.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 66 pat. with knee arthrosocpy
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pain | 24h

SECONDARY OUTCOMES:
Pain drugs | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lierz, MD, Study Chair — Marienkrankenhaus Soest
Locations (1):
- Marienkrankenhaus, Soest, Germany